#### The GlaxoSmithKline group of companies

**Division:** Worldwide Development **Retention Category:** GRS019

**Information Type:** Clinical Reporting and Analysis Plan

| Title: | Clinical Pharmacology Reporting and Analysis Plan for MRI201137: An evaluation of DCE-MRI measures of pulmonary oedema and vascular permeability in healthy subjects and in patients with cardiac failure: A methods validation study for evaluation of novel treatments limiting pulmonary oedema in cardiac failure |
|---|---|
| Compound Number: | GSK2798745 |
| Effective Date: | 28-APR-2017 |

#### **Description**:

The purpose of this reporting and analysis plan (RAP) is to describe the planned analyses and output to be included in the Clinical Pharmacology Study Report for Protocol MRI201137. This RAP is intended to describe the analyses required to validate the use of DCE-MRI for evaluating measures of pulmonary oedema in patients with cardiac failure. This document will be provided to the study team members to convey the content of the final Statistical Analysis Complete (SAC) deliverable.

**Subject:** MRI, heart failure, pulmonary oedema

#### **Author's Name and Functional Area:**

| PPD Lead Statistician | |
|-----------------------|--------------------------------------|
| PPD | Reviewer Statistician |
| PPD | Statistician (simplification of RAP) |

#### Approved via Email by:

The Discovery Biometrics Director (or designee) will give final approval

| PPD | Qsci, Clinical Statistics | 28-APR-2017 |
|-----|---------------------------|-------------|
|-----|---------------------------|-------------|

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

### **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| LIS | T OF A | BBREVIATIONS | 5 |
| 1. | INTRO | DDUCTION | 6 |
| 2. | STUD | Y OBJECTIVE(S) AND ENDPOINT(S) | <mark>7</mark> |
| | 2.1. | Study Objective(s) | 7 |
| 3. | STUD | Y DESIGN | 9 |
| 4. | PLAN | NED ANALYSES | 9 |
| | 4.1. | Interim Analyses | |
| | 4.2. | Final Analyses | 10 |
| 5. | ANAL`<br>5.1. | YSIS POPULATIONSAnalysis Datasets | |
| 6. | | TMENT AND OTHER SUB-GROUP DESCRIPTIONS FOR DATA AYS | 12 |
| 7. | | RAL CONSIDERATIONS FOR DATA ANALYSES AND HANDLING. Reporting Conventions | 12 |
| | 7.2. | Data Management | |
| | 7.3. | Premature Withdrawal and Missing Data | |
| | | 7.3.1. Missing MRI measurements | |
| | 7.4. | 7.3.2. Missing dyspnoea score and respiratory rate | |
| | 7.4.<br>7.5. | Baseline Definition Derived and Transformed Data | |
| | 7.5. | 7.5.1. Change from Baseline | |
| | 7.6. | Values of Potential Clinical Importance | |
| | | 7.6.1. Values of Potential Clinical Importance for Healthy Volunteers | 1/ |
| | | 7.6.2. Laboratory Values of Potential Clinical Importance for | |
| | | Heart Failure Patients | 17 |
| 8. | | Y POPULATION | |
| | 8.1. | Disposition | |
| | 8.2. | Demographic and Baseline Characteristics | 20 |
| 9. | | TY ANALYSES | |
| | 9.1. | Statistical Analyses | |
| | | 9.1.1. Extent of Exposure | |
| | | 9.1.2. Adverse Events | |
| | | 9.1.4. Pregnancies (as applicable) | |
| | | 9.1.5. Clinical Laboratory Evaluations | |
| | 9.2. | Other Safety Measures | |
| | J | 9.2.1. Vital Signs | |
| | | 9.2.2. Respiratory rate | |
| | | 9.2.3. Dyspnoea score | |

#### CONFIDENTIAL

| | | 9.2.4. | ECG Find | ings | 24 |
|---|---|---|---|---|---|
| 10. | | | | | |
| | 10.1. | | | | |
| | | | | and post exercise Analysis | |
| | 10.2. | | | es | |
| | 10.3. | | | S | |
| | | 10.3.1. | | y analyses on other MRI scan measurements | 26 |
| | | 10.3.2. | | on of DLco/DLno parameters at baseline by | |
| | | | group (HV | ', HF) | 27 |
| | | 10.3.3. | Comparis | on of effect of exercise at Scan 3 by group (HV, | |
| | | 4004 | | | 27 |
| | | 10.3.4. | | on of exercise test parameters at Scan 3 by | |
| | | 400= | | <sup>′</sup> , HF) | 27 |
| | | 10.3.5. | Relations | nip between change from baseline MRI scan | |
| | | | | ndpoint (Ve, Ktrans) and change from baseline | |
| | | 4000 | | BNP, DLco/DLno and Ve/VCo2 | |
| | | 10.3.6. | Analysis o | of Group 3 patients | 28 |
| 11. | REFE | RENCES | | | 29 |
| 12. | ATTA | | | | |
| | 12.1. | | Contents for | or Data Display Specifications | 30 |
| | 12.2. | , | | nd Disposition | |
| | | | | ulation | |
| | | 12.2.2. | | n | |
| | | | • • | bhy and Baseline Characteristics | |
| | 12.3. | • | | | |
| | | 12.3.1. | • | to MRI | |
| | | 12.3.2. | | y Data | |
| | 12.4. | | , | | |
| | | 12.4.1. | | 3 | |
| | | 12.4.2. | | | |
| | 12.5. | • | | | |
| | | | | ndpoint | |
| | | | | y endpoint | |
| | | 12.5.3. | | y endpoint | 38 |
| | | | 12.5.3.1. | Exploratory analysis of DCE-MRI | |
| | | | | measurements: Plasma volume (v <sub>p</sub> ), T <sub>1</sub> | 00 |
| | | | 40 5 0 0 | relaxation rate, proton density | 38 |
| | | | 12.5.3.2. | | 4.4 |
| | | | 40 5 0 0 | parameters at baseline by group (HF, HV) | 41 |
| | | | 12.5.3.3. | Comparison of Dyspnoea Score at baseline by group (HV, HF) | 42 |
| | | | 12.5.3.4. | Comparison of Respiratory Rate at baseline by | |
| | | | | group (HV, HF) | 43 |
| | | | 12.5.3.5. | Comparison of effect of exercise at Scan 3 by | |
| | | | | group (HV, HF) | 43 |
| | | | 12.5.3.6. | Comparison of exercise test parameters at | |
| | | | | Scan 3 by group (HV, HF) | 44 |
| | | | | · · | |

#### CONFIDENTIAL

| | 12.5.3.7. | Relationship between exercise parameters (Ve/Vco2) vs gas diffusion DLno/DLco | |
|---|---|---|---|
| | | parameters at scan 3 | 45 |
| 12.6. | Data Display Specif | ications (Example Shells) | 46 |
| - | | | |

## **LIST OF ABBREVIATIONS**

| AE | Adverse Event |
|-----------------|----------------------------------------------------|
| ALT | Alanine Transaminase |
| ANCOVA | Analysis of Covariance |
| AST | Aspartate Transaminase |
| BMI | Body Mass Index |
| BNP | B-Type Natriuretic Peptide |
| CDF | Cumulative Distribution Function |
| DCE | Dynamic Contrast Enhanced |
| DLCO | Diffusing Capacity of the Lung for Carbon Monoxide |
| DLNO | Diffusing Capacity of the Lung for Nitrous Oxide |
| ECG | Electrocardiogram |
| eGFR | Estimated Glomerular Filtration Rate |
| FENa | Fractional excretion of sodium |
| GSK | GlaxoSmithKline |
| HF | Heart Failure |
| HV | Healthy Volunteers |
| ICH | International Conference on Harmonisation |
| Kg | Kilogram |
| Ktrans | Exchange Rate |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mL | Milliliter |
| MRI | Magnetic Resonance Imaging |
| NO | Nitric Oxide |
| NT-proBNP | N-terminal of pro-Brain-type Natriuretic Peptide |
| NYHA | New York Heart Association |
| RAP | Reporting and Analysis Plan |
| RBC | Red Blood Cells |
| RER | Respiratory Exchange Ratio |
| RPE | Rating of Perceived Exertion |
| SAE | Serious Adverse Event |
| SPM | Study Procedures Manual |
| TRPV4 | Transient Receptor Potential Vanilloid 4 |
| $VCO_2$ | Volume of Carbon Dioxide |
| Ve | Interstitial Volume |
| VO <sub>2</sub> | Volume of Oxygen |
| Vp | Plasma Volume |
| WBC | White Blood Cells |

### **Trademark Information**

| Traden | narks of the GlaxoSmithKline group of companies |
|--------|-------------------------------------------------|
| NONE | |

| Trademarks not owned by the GlaxoSmithKline group of companies |
|----------------------------------------------------------------|
| SAS |

### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Pharmacology Study Report for Protocol MRI201137.

| Revision Chronology: | | |
|---|---|---|
| 2013N186309_00 | 2014-FEB-04 | Original |
| 2013N186309_01 | 2014-APR-24 | Amendment No.: 01 This protocol amendment clarifies the exercise protocol to be conducted, details measures for endpoints, defines the biomarker to be measured (NT-pro BNP), reduces total blood volume to be collected, updates study schematic, adds an interim review of the data, removes collection of AEs as there is no IP included in the study, alters physical exams to brief physical exams, and adds a dyspnoea scale and the Borg Rating of Perceived Exertion. |
| 2013N186309_02 | 2015-FEB-16 | Amendment No.: 02 This protocol amendment changes modifies inclusion criteria, clarifies the exercise protocol, and corrects the footnote numbering in the time and events table. |
| 2013N186309_03 | 2016-APR-08 | Amendment No. 3 adds an evaluation of an additional group of subjects who have been hospitalized for acute decompensated heart failure to determine whether DCE-MRI can detect changes in measures of pulmonary oedema with standard of care treatment. Details for summarizing data from ADHF patients (referred to in this document as group 3) can be found in Section 10.2.6. |
| 2013N186309_03 | 2016-APR-20 | The data analysis for Group 3 has been simplified due to limited number of subjects (n=3) in the study |

In addition to following the revision chronology of the study protocol, current reversions are also under the general guidance of "driving efficiency in Clinical Statistics" initiative,

and the outputs are simplified to match with the scale and lack of investigational drug of the study.

All decisions regarding final analysis, as defined in this RAP document, have been made prior to Database Freeze of the study data. After completion of 12 evaluable subjects, an informal interim look will be performed.

## 2. STUDY OBJECTIVE(S) AND ENDPOINT(S)

### 2.1. Study Objective(s)

The objectives and endpoints for the study are summarized in the table below:

| | Objectives | Endpoints | |
|---|---|---|---|
| Pri | mary | • | |
| • | Establish whether DCE-MRI can detect differences in measures of pulmonary oedema or vascular permeability between HF and healthy volunteers (HV) groups. | • | Interstitial volume (ve) and exchange rate (ktrans) measured using DCE-MRI in HF patients and HVs at baseline. |
| • | Explore the effect of exercise on DCE-MRI measures of pulmonary oedema and vascular permeability in HF and HV groups. | • | Change in interstitial volume (ve) and exchange rate (ktrans) measured using DCE-MRI in HF patients and HVs before and following exercise. |
| • | Explore the effect of standard of care treatment on DCE-MRI measures of pulmonary oedema and vascular permeability in patients with ADHF. | • | Change in interstitial volume (ve) and exchange rate (ktrans) measured using DCE-MRI in patients with ADHF during hospitalization and following the resolution of pulmonary oedema. |
| Sec | condary | | |
| • | Estimate the intra subject variability of DCE-MRI measures of pulmonary oedema and vascular permeability. | • | Estimation of the variability in the interstitial volume (ve) and exchange rate (ktrans) within HF patients and HVs between 2 MRI visits approximately 1 week apart. |

| Objectives | Endpoints |
|---|---|
| Exploratory | |
| Explore the relationship between DCE-MRI measures of pulmonary physiology and disease severity, symptoms, pulmonary function, volume status and renal function | Correlation of MRI measures with clinical and biochemical measures: dyspnoea score, respiratory rate, NT-proBNP, exercise capacity (including BORG RPE, heart rate, blood pressure and gas exchange endpoints such as peak VO2, Ve/VCO2 slope), DLCO, DLNO, body weight, urine specific gravity, fractional excretion of sodium (FENa), blood urea to creatinine ratio. |
| Estimate differences in plasma volume<br>and MR physical properties<br>influenced by the tissue<br>microenvironment relaxation rate, and<br>proton density between HF and HV<br>groups as measured using DCE-MRI | Plasma volume (vp), T1 relaxation rate, and proton density measured using MRI in HF patients and HVs. |
| Explore the distribution of DCE-MRI measures of pulmonary physiology in HF and HV groups both before and after exercise | • Interstitial volume (ve) and exchange rate (ktrans), and other clinical and biochemical measures as listed above if data permit. |
| • Explore the effect of standard of care treatment on plasma volume and MRI physical properties influenced by the tissue microenvironment relaxation rate, and proton density in patients with ADHF. | • Change in Plasma volume (vp), T1 relaxation rate, and proton density measured using MRI in patients with ADHF during hospitalization and following the resolution of pulmonary oedema; |
| Explore the effect of standard of care treatment on ultrasound measures of pulmonary oedema in patients with ADHF. | Change in B-lines measured using ultrasound in patients with ADHF during hospitalization and following the resolution of pulmonary oedema; |
| • Explore the distribution of DCE-MRI measures of pulmonary physiology in ADHF patients both before and after standard of care treatment; | Interstitial volume (ve) and exchange rate (ktrans), and other clinical and biochemical measuresas listed above if data permit; |

#### 3. STUDY DESIGN

The study will enroll 12 HV and 12 HF patients. First, the DCE-MRI markers of vascular permeability and pulmonary edema will be measured in HV and HF patients at rest to determine whether there is a difference between the two populations. Next, exercise-induced changes relative to rest in interstitial volume and exchange rate will be evaluated in both HV and HF patients. Since exercise increases pulmonary vascular pressure more markedly in patients with left ventricular failure as compared to normal subjects, a greater increase in vascular permeability and pulmonary oedema may be observed in patients with HF as compared to HV.

The study consists of four visits. The first visit will be a Screening Visit during which the subjects will be assessed for their tolerance of lying flat and baseline information will be collected. Within 35 days, subjects will return for the first of two scanning sessions approximately one week apart to determine baseline levels and within subject variability. A third imaging visit will incorporate a bicycle exercise challenge prior to imaging and will occur approximately one to three days after the second imaging session.

All MRI data will be anonymized at site and transferred to Bioxydyn Limited for DCE-MRI data analysis. The 'extended Tofts' tracer kinetic model will be applied to the data to provide measurements of  $k^{\text{trans}}$  (capillary transfer coefficient of contrast agent - /min),  $v_e$  (leakage space - fraction) and  $v_p$  (plasma volume - fraction). Median values of  $k^{\text{trans}}$  and  $v_e$  will be provided from each lung (total lung, apical and basal) as well as total lung for subsequent statistical analysis. All values will be corrected for the individual's hematocrit value. If not available, a typical hematocrit value will be assumed.

In Session 3 (which will be conducted in 2 visits), subjects will perform two exercise tests. Subjects will first be asked to perform a maximal exercise test limited by dyspnoea or fatigue on a cycle ergometer. At the 2nd visit, subjects will be asked to perform cycle exercise for 10 minutes at 75%-80% of the peak work rate achieved during the maximal exercise to exhaustion test described above.

For subjects with ADHF (Group 3), the study design is shown below:



#### 4. PLANNED ANALYSES

### 4.1. Interim Analyses

After 12 evaluable subjects (6 HV and 6 HF patients) have completed Sessions 1 and 2, an interim review will be performed. Following the interim review, the study team will decide whether to (a) terminate the study if it is determined that the image quality is poor

(e.g., due to excessive movement during scanning or related to specifics around lung tissue) or the procedures are not well tolerated in the HF group (e.g., inability to lie flat for the duration of the imaging session), or (b) continue the study and enrol an additional 12 evaluable subjects (6 HV and 6 HF patients).

The interim decision will be based on the expert opinion of the Investigator in consultation with the GSK Study Team based on the totality of the data. No formal interim analysis will be reported out.

#### 4.2. Final Analyses

The final planned analyses will be performed after all subjects have completed the study and after database freeze. See Section 9 to Section 10 for all final planned analyses for this study.

#### 5. ANALYSIS POPULATIONS

An evaluable subject is defined as a subject that has MRI data of sufficient quality to enable DCE-MRI modelling in both Session 1 and Session 2.

#### All enrolled population

The all enrolled population will include all subjects who have signed the informed consent for participation in the study.

#### Safety population

The safety population will include all enrolled subjects who have initiated Session 1 DCE-MRI scan. All safety analyses will be based on the safety population.

For Group 3, the safety population will include all enrolled subjects who have initiated at least one session of DCE-MRI or LUS scan.

This is the population to be used for all tables, listings, and figures of patients in group 3.

#### **Evaluable** population

The evaluable population will include subjects in safety population who are 40 years and older .There is no plan to exclude subjects with major or minor protocol deviations from the analyses. However, subject data will be examined for evidence of protocol deviations in order to assess how well the protocol was followed. If necessary, any decision to exclude any subject from the planned analyses will be determined when the database is released for reporting purposes.

The evaluable populations have been changed in this RAP amendment to limit the analysis populations to subjects with age greater than 40 years old at baseline. At the interim analysis, it was realized that age may confound the results in the HV population. Since HV and HF subjects were not age-matched, limiting the analysis population to similar age range will provide a more appropriate comparison. This analysis will exclude

4 subjects; however, the study has enrolled an additional 5 subjects who are >40 years old in order to have a sufficient number of subjects for comparison. However, in addition to the comparisons using the defined populations in this RAP, a sensitivity analysis for the comparison between two groups on the change from baseline in Ve will be performed using safety population with all subjects who have evaluable MRI data in either Sessions 1 or 2.

The evaluable population definition does not apply to ADHF patients to be included in in group 3 summaries.

This population is not applicable to Group 3.

#### 5.1. Analysis Datasets

#### **Primary Analysis Set**

The primary analysis set to evaluate whether DCE-MRI can detect differences in measures of pulmonary oedema or vascular permeability between HV and HF patients will include all subjects in the evaluable population. A sensitivity analysis for Ve will also be performed using the safety population.

This analysis set will also be used to explore the effect of exercise on DCE-MRI measures in HV and HF patients. Missing post-exercise MRI data will not be imputed. This analysis set will be used to estimate the intra-subject variability of DCE-MRI measures of pulmonary oedema and vascular permeability.

#### **Secondary Analysis Set**

The secondary analysis set will include all evaluable subjects who have MRI data of sufficient quality from Session 1, 2 or both. This analysis set will be used to estimate the intra-subject variability of DCE-MRI measures of pulmonary oedema and vascular permeability.

No formal hypothesis testing will be performed.

No analysis will be performed for Group 3, so no analysis data sets will be defined.

# 6. TREATMENT AND OTHER SUB-GROUP DESCRIPTIONS FOR DATA DISPLAYS

| Population Group | | Final Data Display (i.e. HARP / other) Treatment Description |
|---|---|---|
| Code Treatment Description | | Treatment Description |
| HV | Healthy Volunteer | Healthy Volunteer |
| HF | Heart Failure Patient | Heart Failure Patient |
| ADHF | Acute Decompensated Heart Failure | Acute Decompensated Heart Failure Patient |

# 7. GENERAL CONSIDERATIONS FOR DATA ANALYSES AND HANDLING

### 7.1. Reporting Conventions

Data manipulations and statistical analyses will be performed using SAS version 9.2 or higher.

All variables will be presented and summarized in tables or graphs. Continuous variables will be summarized using descriptive statistics (mean, standard deviation, median, interquartile range (where appropriate), and range). Categorical variables will be summarized using frequency counts and percentages. Associated listings will also be provided. Unless otherwise stated, 95% confidence intervals around the point estimates, as appropriate will be presented.

### 7.2. Data Management

| Data Type | Source | Format of Data | Planned Date of Final File <sup>1</sup> | Responsibility |
|---|---|---|---|---|
| Safety | Database | IDSL | DBF | CPSSO |
| PD/biomarker | Study Site | CSV file | DBF | CPSSO |

<sup>1.</sup> This is for study teams to determine upfront if there is a possibility of not meeting the completion of the CPSR within 6 months of LSLV (i.e. novel data that may not be available until several months after LSLV).

## 7.3. Premature Withdrawal and Missing Data

All subjects who withdraw prematurely from the study will be documented and the reason for their withdrawal recorded in the final Clinical Pharmacology Study Report (CPSR). All available data from subjects who withdraw will be listed and all available planned data will be included in the summaries according to the populations and analysis datasets defined in Section 5.

#### 7.3.1. Missing MRI measurements

Session 1 and Session 2 MRI measurements can be considered baseline pre-exercise data. If Session 2 data is unavailable, Session 1 data will be used. For the purpose of the secondary analysis to estimate intra-subject variability, MRI data will not be imputed.

#### 7.3.2. Missing dyspnoea score and respiratory rate

The last available dyspnoea score or respiratory rate will be carried forward in the case of missing Session 2, and pre-exercise Session 3 measurements. Post-exercise measurements will not be imputed.

Other missing data will not be imputed.

#### 7.4. Baseline Definition

The Session 2 visit will be considered as the baseline visit for MRI measurement endpoints. If Session 2 data is unavailable, Session 1 data will be used. In terms of change from baseline calculation for statistical analysis, tables below defined the baseline for each endpoint of interests:

| | | Baseline Colle | Baseline To Be Used in Analysis / Summaries | |
|---|---|---|---|---|
| | Screening | Session 2/1 | | |
| Parameter | | | | |
| MRI scan | | Χ | Х | Scan 2 |

Note: For the parameters of MRI scan, if measurements are missing for Scan 2, then Scan 1 measurements will be used as baseline.

| | | Baseline Coll | Baseline To Be Used in Analysis / Summaries | |
|---|---|---|---|---|
| | Screening | Session 2/1 | Session 3 | |
| Parameter | | | | |
| Laboratory | Х | | Pre-Excercise | Session 3 Pre- |
| biomarker | _ ^ | | Pre-Excercise | Excercise |
| Dooniratory rata | | Post-MRI | Pre-Excercise | Session 3 Pre- |
| Respiratory rate | | PUSI-IVIRI | Fie-Excercise | Excercise |
| Dyspnoea Scale | | Doot MDI | Dro Eventoine | Session 3 Pre- |
| Scoring | | Post-MRI | Pre-Excercise | Excercise |
| Gas Diffusion, | | Doot MDI | Dro Evocacion | Session 3 Pre- |
| DL <sub>co</sub> , DL <sub>no</sub> | | Post-MRI Pre-Excercise | | Excercise |
| Pulmonary | | Doot MDI Dro Evecroine | | Session 3 Pre- |
| function | | Post-MRI | Pre-Excercise | Excercise |

#### 7.5. Derived and Transformed Data

MRI measures: Median values of  $k^{\text{trans}}$ ,  $v_e$  and  $v_p$  from multiple images/regions will be calculated for total lung, each lung (left and right) and different lung segments. For each MRI measure parameter there are 7 measurement regions: total lung, left lung, right lung, apical left segment, apical right segment, basal left segment and basal right segment for each MRI measure parameter.

Laboratory Data: The majority of laboratory results will be recorded under a numeric field. Some results may be recorded under a character field where a numeric component

(x) has been preceded by '>' or '<' indicating the true value of x is greater than or less than that given.

To ensure this data is not excluded from any summaries or analysis, any laboratory results recorded as '>x' will be moved to the numeric field with a value of x, similarly results recorded as '<x' will be moved to the numeric field with a value of x. All listings will present the data as recorded.

*Age (years):* Age will be calculated using the date of the screening visit relative to year of birth, according to the Integrated Data Standard Library (IDSL). In this calculation, date of birth will be imputed based on the assumption that all subjects were born on the 30<sup>th</sup> June (30 Jun YYYY).

Body Mass Index (BMI)  $(kg/m^2)$ : equals (weight (kg)) / ((height (m))<sup>2</sup>)

Study Day: Study day will be defined in reference to the DCE-MRI scan date in the corresponding Session. Session 1 – Day 1 will be the DCE-MRI scan date in Session 1, and Session 2 – Day 1 will be the DCE-MRI scan date in Session 2, etc.

#### 7.5.1. Change from Baseline

The change from baseline will be calculated by subtracting the baseline values from the individual post-exercise values. If either the baseline or post-exercise value is missing, the change from baseline is set to missing as well.

## 7.6. Values of Potential Clinical Importance

#### 7.6.1. Values of Potential Clinical Importance for Healthy Volunteers

| Hematology Analyte | Effect | Relative – Low<br>(Multipliers of LLN) | Relative – High<br>(Multipliers of ULN) |
|---|---|---|---|
| White Blood Cell Count | | 0.67 | 1.82 |
| Neutrophil Count | | 0.83 | |
| Hemoglobin | Male | | 1.03 |
| | Female | | 1.13 |
| Hematocrit | Male | | 1.02 |
| Hematocrit | Female | | 1.17 |
| Platelet Count | | 0.67 | 1.57 |
| Lymphocytes | | 0.81 | |

| Chemistry Analyte | Effect | Relative – Low<br>(Multipliers of LLN) | Relative – High<br>(Multipliers of ULN) |
|---|---|---|---|
| Albumin (mmol/L) | | 0.86 | |
| Calcium (mmol/L) | | 0.91 | 1.06 |
| Glucose (mmol/L) | | 0.71 | 1.41 |
| Magnesium (mmol/L) | | 0.63 | 1.03 |
| Phosphorus (mmol/L) | | 0.80 | 1.14 |
| Potassium (mmol/L) | | 0.86 | 1.10 |
| Sodium (mmol/L) | | 0.96 | 1.03 |
| Total CO <sub>2</sub> (mmol/L) | | 0.86 | 1.14 |

# **Liver Function Test (Healthy Volunteers)**

| <b>Liver Function Test</b> | Effect | Potential Clinical Importance (PCI) | Unit |
|---|---|---|---|
| Analyte | Effect | Range | |
| ALT/SGPT | High | $\geq 2x \text{ ULN}$ | U/L |
| AST/SGOT | High | $\geq 2x \text{ ULN}$ | U/L |
| AlkPhos | High | $\geq 2x \text{ ULN}$ | U/L |
| T. Bilirubin | High | ≥ 1.5x ULN | μmol/L |
| | | ≥ 1.5x ULN T.Billirubin | μmol/L |
| T. Bilirubin + ALT | High | + | |
| | | $\geq 2x$ ULN ALT | U/L |

# **ECG Values of Potential Clinical Importance (Healthy Volunteers)**

| ECG Parameter | Potential Clinical Importance<br>Range (PCI) | Unit |
|---|---|---|
| Absolute QTc Interval | >450 | msec |
| Increase from Baseline QTc | >60 | msec |
| PR Interval | <110 and >220 | msec |
| QRS Interval | <75 and >110 | msec |

| ECG Parameter | Potential Clinical Importance Range (PCI) | Unit |
|---|---|---|
| Absolute QTc Interval | >450 to <480 | msec |
| Absolute QTc Interval | >480 to \le 500 | msec |
| Absolute QTc Interval | >500 | msec |
| Increase from Baseline QTc | >30 to ≤60 | msec |
| Increase from Baseline QTc | >60 | msec |

## **Vital Sign Values of Potential Clinical Importance (Healthy Volunteers)**

| VS Parameter | Potential Clinical Importance Range (PCI) | Unit |
|--------------------------|-------------------------------------------|------|
| Systolic Blood Pressure | <85 and >160 | mmHg |
| Diastolic Blood Pressure | <45 and >100 | mmHg |
| Heart Rate | <40 and >110 | bpm |

## **Vital Sign Values of Potential Clinical Importance (Healthy Volunteers)**

| VS Parameter | Potential Clinical Importance Range (PCI) | Unit |
|--------------------------|-------------------------------------------|------|
| Systolic Blood Pressure | Increase $\geq 20$ and $\geq 40$ | mmUa |
| (Change from Baseline) | Decrease $\geq 20$ and $\geq 40$ | mmHg |
| Diastolic Blood Pressure | Increase $\geq 10$ and $\geq 20$ | mmUa |
| (Change from Baseline) | Decrease $\geq 10$ and $\geq 20$ | mmHg |
| Heart Rate | Increase $\geq 15$ and $\geq 30$ | hom |
| (Change from Baseline) | Decrease $\geq 15$ and $\geq 30$ | bpm |

# 7.6.2. Laboratory Values of Potential Clinical Importance for Heart Failure Patients

Note GI/L =  $10^9/L=10^3/\mu L$ 

| Hematology | | | |
|---|---|---|---|
| Laboratory<br>Test | Units | Change from Baseline of<br>Potential Clinical<br>Concern | Potential Clinical<br>Concern Value |
| Basophils | GI/L | None | None |
| Calcitonin | pg/mL | None | >100 pg/mL |
| Eosinophils | GI/L | None | None |
| Hematocrit | 1 | >0.1 decrease | >0.05 below LLN<br>>0.04 above ULN |
| Hemoglobin | g/L | >25 g/L decrease | >20 g/L below LLN<br>>10 g/L above ULN |
| Lymphocytes | GI/L | None | <0.5 x LLN |
| Monocytes | GI/L | None | None |
| Neutrophils | GI/L | None | <1 GI/L |
| Platelet<br>Count | GI/L | None | <80 GI/L<br>>500 GI/L |
| Red Blood<br>Cell Count | TI/L | None | None |
| White Blood<br>Cell Count | GI/L | None | >1 GI/L below LLN<br>>5 GI/L above ULN |

| | Chemistry | | |
|---|---|---|---|
| Laboratory<br>Test | Units | Change from Baseline of<br>Potential Clinical<br>Concern | Potential Clinical<br>Concern Value |
| Albumin | g/L | None | None |
| Alkaline<br>Phosphatase | U/L | None | >3 x ULN |
| ALT | U/L | None | >3 x ULN |
| AST | U/L | None | >3 x ULN |
| Bicarbonate<br>(Carbon<br>Dioxide | mmol/L | None | <16 mmol/L > 40 mmol/L |

| | Chemistry | | |
|---|---|---|---|
| Laboratory<br>Test | Units | Change from Baseline of<br>Potential Clinical<br>Concern | Potential Clinical<br>Concern Value |
| Content) | | | |
| Blood Urea<br>Nitrogen | mmol/L | None | >2 x ULN |
| Calcium | mmol/L | None | <1.8 mmol/L<br>>3.0 mmol/L |
| Chloride | mmol/L | None | None |
| Creatinine | umol/L | ≥50% increase from baseline | >159 umol/L |
| Direct<br>Bilirubin | umol/L | None | >1.35 x ULN |
| Gamma<br>Glutamyl<br>Transferase | U/L | None | >3 x ULN |
| Glucose (fasting) | mmol/L | None | <3 mmol/L<br>>22 mmol/L |
| Magnesium | meq/L | None | ≤1 meq/L |
| Potassium | mmol/L | None | >0.5 mmol/L below<br>LLN<br>>1.0 mmol/L above<br>ULN |
| Sodium | mmol/L | None | >5 mmol/L above LN or below LN |
| Total<br>Bilirubin | umol/L | None | >1.5 x ULN |
| Total Protein | g/L | None | >15 g/L above or below LN |
| Uric acid | umol/L | None | >654 umol/L |

| Liver Function Test | |
|---|---|
| <b>Laboratory Test</b> | Potential Clinical Concern Value |
| ALT | ≥2 x ULN |
| | $\geq$ 3 x ULN |
| | $\geq$ 5 x ULN |
| | $\geq$ 8 x ULN |
| | $\geq$ 10 x ULN |
| | $\geq$ 3 x ULN and Total Bilirubin $\geq$ 2 x ULN |
| AST | ≥2 x ULN |
| | $\geq$ 3 x ULN |
| | $\geq$ 5 x ULN |
| | ≥8 x ULN |
| | $\geq$ 10 x ULN |
| | $\geq$ 3 x ULN and Total Bilirubin $\geq$ 2 x |
| | ULN |
| Total Bilirubin | ≥ 1.5 x ULN |
| | $\geq$ 2 x ULN |
| | $\geq$ 3 x ULN |
| | ≥ 5 x ULN |
| | ≥8 x ULN |
| | ≥ 10 x ULN |

# **Vital Signs**

| Parameter | Units | Change from Baseline of<br>Potential Clinical Concern | Potential Clinical<br>Concern Value |
|---|---|---|---|
| Systolic BP | mmHg | Decrease >30 mmHg<br>Increase >30 mmHg | <100 mmHg<br>>170 mmHg |
| Diastolic BP | mmHg | Decrease >20 mmHg Increase >20 mmHg | <50 mmHg<br>>110 mmHg |
| Heart rate | bpm | Decrease >30 bpm<br>Increase >30 bpm | <50 bpm<br>> 120 bpm |

#### **ECG**

| Parameter | Units | Change from Baseline of Potential<br>Clinical Concern | Potential<br>Clinical<br>Concern Value |
|---|---|---|---|
| Heart Rate | bpm | Decrease >30 bpm<br>Increase >30 bpm | Supine: < 50 or > 120 bpm |
| QRS interval | msec | Increase of > 25% when baseline QRS >100 msec Increase of > 50% when baseline QRS ≤100 msec | >200 msec |
| QTcB | msec | Increase of > 10% when baseline QTc >440 msec Increase of > 20% when baseline QTc ≤440 msec | >500 msec |
| QTcF | msec | Increase of > 10% when baseline QTc >440 msec Increase of > 20% when baseline QTc <440 msec | >500 msec |
| PR Interval | msec | Increase of > 25% when baseline PR >200 msec Increase of > 50% when baseline PR <200 msec | >300 msec |

#### 8. STUDY POPULATION

The precise format and content of the Study Population tables are shown in Section 12.2 of the RAP.

### 8.1. Disposition

Data displays will be produced to account for all subjects enrolled in the study. This will include the number of subjects enrolled in each population (HV or HF patients), number of subjects who have attempted or completed the DCE-MRI scan at each session, number of early withdrawals and reasons for early withdrawal. Number of subjects in each analysis population as defined in Section 5 will also be summarized.

The tables will use the "All subjects" population unless otherwise specified.

## 8.2. Demographic and Baseline Characteristics

Demography data will be summarized for safety population in this study. Disease characteristics data will also be summarized for the HF patients if data are available

These will include the following:

• Year of birth

- Gender
- Race and ethnicity
- Significant past medical history including onset, aetiology, and results of any recent relevant investigations of heart failure, as applicable
- Medication history
- Confirm heart failure class (HF patients only)
- Onset and type of symptoms (HF patients only)
- Years since diagnosis of HF (HF patients only)
- Degree of exercise intolerance-- distance/ stairs/time prior to breathlessness
- Presence of orthopnoea and/or paroxysmal nocturnal dyspnoea
- Peripheral oedema—level above ankle, non-dependent limb

#### 9. SAFETY ANALYSES

The precise format and content of Safety figures, tables and listings are shown in Section 12.3 of the RAP.

The tables will use the "Safety" population unless otherwise specified.

#### 9.1. Statistical Analyses

#### 9.1.1. Extent of Exposure

No treatment (investigational product) will be given in this study. The number of subjects who were exposed to 1 MRI scan, 2 MRI scans, or 3 MRI scans will be summarized. Subjects who completed scan 1 and scan 2, but could not complete scan 3, with reason will be listed. If more than one patient cannot complete scan 3 due to not being able to lie down, an additional exploratory analysis will be undertaken.

#### 9.1.2. Adverse Events

Since no investigational product will be administered in this study, information regarding the occurrence of adverse events will not be routinely collected. Medical occurrences (non-serious events) that begin during the study may be recorded under Medical History/Current Medical Conditions. Non-serious events related to study procedures may also be recorded.

Any SAEs assessed as related to study participation (e.g., protocol-mandated procedures, invasive tests, or change in existing therapy) will be recorded from the time a subject consents to participate in the study up to and including the last visit.

Any SAEs assessed as related to study procedures will be recorded. SAEs will be coded and grouped by system organ class (SOC) and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA).

Based on date/time of onset, session number will be assigned to each SAE and duration from last MRI scan will be calculated.

| Session | Definition |
|---------|----------------------------------------------------|
| 0 | AEs with onset prior to Session 1 MRI |
| 1 | AEs with onset between Session 1 and Session 2 MRI |
| 2 | AEs with onset between Session 2 and Session 3 MRI |
| 3 | AEs with onset after Session 3 MRI |

Frequency of SAEs will be summarized by subject population overall and by session. A SAE will only be counted once within a session.

#### 9.1.3. Deaths and Serious Adverse Events

Deaths, as well as SAEs, if any, leading to discontinuation of the study will be presented in separate listings

### 9.1.4. Pregnancies (as applicable)

Any pregnancies reported or identified during this study will be listed.

#### 9.1.5. Clinical Laboratory Evaluations

Haematology, clinical chemistry, urinalysis and additional parameters to be tested are listed below. Baseline clinical laboratory data will be collected for all HV and HF patients. Additional laboratory data will be collected before the MRI scan at each session for the HF patients.

Haematology

| Platelet Count | Automated WBC Differential: |
|----------------------|-----------------------------|
| RBC Count | Neutrophils |
| WBC Count (absolute) | Lymphocytes |
| Hemoglobin | Monocytes |
| Hematocrit | Eosinophils |
| | Basophils |

#### **Clinical Chemistry**

| Urea | Potassium | Total and direct bilirubin |
|------------|------------|---------------------------------------|
| Creatinine | Troponin | eGFR (estimated Glomerular Filtration |
| | | Rate) |
| Glucose | Calcium | |
| Sodium | AST (SGOT) | |
| Potassium | ALT (SGPT) | |

#### **Routine Urinalysis**

| V |
|-----------------------------------------------------------|
| Specific gravity |
| pH, glucose, protein, blood and ketone by dipstick |
| Microscopic examination (if blood or protein is abnormal) |

#### **Biomarkers**

N-terminal pro-Brain-type Natriuretic Peptide (NT- pro BNP)

Descriptive statistics and number of subjects with abnormal clinical laboratory values will be summarized by subject population and by session (in HF patients only).

### 9.2. Other Safety Measures

#### 9.2.1. Vital Signs

Vitals signs, including systolic blood pressure, diastolic blood pressure and heart rate, will be collected at screening, and after MRI scan in Sessions 1 and 2. In Session 3, data will also be collected at the beginning and at the end of the maximal exercise test and the constant workload exercise test. Descriptive statistics for the measurements in all sessions and change from pre-exercise will be provided.

#### 9.2.2. Respiratory rate

Respiratory rate will be collected after MRI scan in Session 1 and Session 2. In Session 3, data will also be collected at the beginning and at the end of the maximal exercise test and the constant workload exercise test. Data will be also collected after MRI scan in constant exercise test. Descriptive statistics for the measurements in all sessions and change from pre-exercise in session 3 will be provided.

#### 9.2.3. Dyspnoea score

Dyspnoea score will be collected after MRI scan in Sessions 1 and 2. In Session 3, data will also be collected before and after the maximal exercise test and the constant workload exercise test. Also data will be collected after MRI scan in constant workload visit. The dyspnoea score data is (0,1,2,3,45), descriptive statistics for the measurements

<sup>\*</sup>At Screening and in Session 3 only, blood samples for NT-Pro BNP determinations will be drawn before and after the maximal exercise test, before the constant workload exercise test and after MRI scanning only in subjects with HF.

in all sessions and change from pre-exercise in session 3 will be provided, in addition a bar chart showing the frequency of each score will be presented.

#### 9.2.4. ECG Findings

12-lead ECGs will be obtained at screening. Results will be displayed in the baseline characteristics table described in Section 9.2.

#### 10. VALIDATION ANALYSES

Planned analyses for the primary, secondary and exploratory objectives of the study are described in this section using the evaluable population as the primary analysis population. Listings of all MRI data, clinical and biochemical measures will be produced. Special listings, such as listings that include data from multiple sources or include only a subset of subjects/measurements are described in the corresponding sections below.

#### 10.1. Primary Objectives

#### 10.1.1. Baseline and post exercise Analysis

For the primary endpoints, contrast agent interstitial volume ( $v_e$ ) and exchange rate ( $k^{trans}$ ) data for total lung, left and right lung, apical segments and basal segments for each lung (total 7 measurements for each parameter) will be fitted separately using a repeat measure ANOVA model with terms include patient population (HF or HV), visit (i.e. sessions), interaction of patient population and visit, with subject ID as block of the repeat factor. Point estimates and associated 95% confidence intervals (CI) will be constructed to provide a plausible range of values for the following parameters of interest: mean DCE-MRI measurements in HV and HF patients, and the mean difference between the HV and HF groups, at each session, as well as the differences among MRI sessions within each patient population group (HV or HF) See example sas codes below.

```
/* analysis of primary endpoints to compare HF vs HV with Sessions 1 to
3 data */
proc mixed data=mri;
  class subjid atrtgrp visit;
 model mriresn = visit atrtgrp visit*atrtgrp/e3 ddfm=kr outp=pred one;
  repeated visit/ subject=subjid type=un;
 by mritstu regint;
 LSMEANS visit*atrtgrp /CL ALPHA=0.05;
  estimate 'HF - HV at Session 1' atrtgrp 1 -1
                      visit*atrtgrp 1 0 0 -1 0 0/cl alpha = 0.05;
   estimate 'HF - HV at Session 2' atrtgrp 1 -1
                      visit*atrtgrp 0 1 0 0 -1 0/cl alpha = 0.05;
   estimate 'HF - HV at post excercise' atrtgrp 1 -1
                      visit*atrtgrp 0 \ 0 \ 1 \ 0 \ 0 \ -1/cl alpha = 0.05;
   estimate 'Session 2 - Session 1 in HF' visit -1 1 0
                      visit*atrtgrp -1 1 0 0 0 0/cl alpha = 0.05;
   estimate 'post excercise - Session 1 in HF' visit -1 0 1
                       visit*atrtgrp -1 0 1 0 0 0/cl alpha = 0.05;
   estimate 'change from baseline estimates in HF' visit 0 -1 1
                       visit*atrtgrp 0 -1 1 0 0 0/cl alpha = 0.05;
```

#### 10.2. Secondary Objectives

For the secondary endpoint, the estimation of the within subject variability of DCE-MRI measures of pulmonary edema and vascular permeability between study visits will be calculated based on the mixed model described in Section 10.1.1, but with Session 1 and 2 data, with log\_e transformation. For the by patient population estimates, a repeated measure ANOVA model will be fitted with visit as the effect effects. The within subject variability (coefficient of variation) can then be estimated as 100\*sqrt(exp(mse)-1), where MSE is the mean square error from the mixed effects model. Example sas codes as follows:

```
/* analysis of primary endpoints to assess variability of primary
endpoints with Sessions 1 to 2 data (secondary endpoint of the analysis
/* estimate overall within subject variability */
data mri Session12;
   set mri;
   if visit in ('SESSION 1' 'SESSION 2');
  if mriresn>0 then lg mriresn=log(mriresn);
proc mixed data=mri Session12;
  class subjid atrtgrp visit;
 model lg mriresn = visit atrtgrp visit*atrtgrp/e3 ddfm=kr
outp=pred one;
 random subjid;
 by mritstu regint;
 ods output covparms = cov one;
 run;
data cvb1;
    set cov one;
      where CovParm="Residual";
  mse=estimate;
 keep mritstu regint mse;
  data cvb2;
     set cov one;
     where CovParm="SUBJID";
 subj=estimate;
 keep mritstu regint subj;
data covp0;
    merge cvb1 cvb2;
```

```
by mritstu regint;
       cvw=compress(put(100*sqrt(exp(mse)-1),5.1));
    keep mritstu regint cvw;
run;
proc sort data=mri Session12;
   by mritstu regint atrtgrp;
/*obtain within subject varibility by patient population */
proc mixed data=mri Session12;
  class subjid atrtgrp visit;
 model lg mriresn = visit /e3 ddfm=kr outp=pred one;
 random subjid;
 by mritstu regint atrtgrp;
 ods output covparms = cov one1;
data cvb11;
     set cov one1;
     where CovParm="Residual";
  mse=estimate;
 keep mritstu regint atrtgrp mse;
  data cvb12;
      set cov one1;
      where CovParm="SUBJID";
 subj=estimate;
 keep mritstu regint atrtgrp subj;
data covp01;
     merge cvb11 cvb12;
       by mritstu regint atrtgrp;
       cvw=compress(put(100*sqrt(exp(mse)-1),5.1));
      keep mritstu regint atrtgrp cvw;
run;
```

### 10.3. Exploratory Analysis

### 10.3.1. Exploratory analyses on other MRI scan measurements

DCE-MRI measurements, including change from baselines, will be summarized by visit. The corresponding mean (SE) plots with separate line for HF and HV will be provided also.

A Spaghetti plot for each parameter, with scan session along the horizontal axes, a line for each subject (differentiate HV and HF by different symbol) representing values for the parameter on the vertical axes, will be provided.

Listings with DCE-MRI measurements will be presented.

The distribution of DCE-MRI measures of pulmonary physiology (interstitial volume  $(v_e)$ , exchange rate  $(k^{trans})$  and Plasma volume  $(v_p)$ ) in HV and HF patients both before and after exercise will be plotted using a scatter plot.

# 10.3.2. Comparison of DLco/DLno parameters at baseline by group (HV, HF)

The similar analysis as for the primary endpoint (Section 10.1.1) will be presented for the parameters of gas diffusion DLco/DLno such as DLNO, DMCO, at baseline and post exercise if data permit.

### 10.3.3. Comparison of effect of exercise at Scan 3 by group (HV, HF)

The analysis will be based on the Evaluable population. The change from baseline parameters of interest on pre-exercise test to post-exercise test in Scan 3 will be fitted separately using a mixed effect model with subject as a random effect, patient population (HF or HV) as fixed effects. Point estimates and associated 95% confidence intervals (CI) will be constructed to provide a plausible range of values for the mean change from baseline measurements in HV and HF patients in Session 3, and the mean difference between the HV and HF groups. Gas diffusion DLco/DLno and lung function parameters in constant exercise session at Scan 3. Change from baseline pre-exercise workload test to post-exercise test is defined as:

DLco/DLno: Scan 3 post MRI – Scan 3 pre-exercise

Lung function: Scan 3 post MRI – Scan 3 pre-exercise

In addition, NT-ProBNP (heart failure patients only), Dyspnoea Score, Respiratory Rate, parameters for gas diffusion and DLco/DLno will be summarized by planned time and group (HV, HF) at Scan 3 by separate exercise session. The corresponding mean (SE) plots will be provided also.

(keep if already programmed)

# 10.3.4. Comparison of exercise test parameters at Scan 3 by group (HV, HF)

The similar analysis as for the primary endpoint (Section 10.3.6) will be presented for exercise test on parameters of interests including Ve/Vco2 ratio at Scan 3 in maximal test and constant exercise session separately. See below for the example sas codes for the analysis:

```
ods output covparms = cov_one;
ods output estimates = est;
run;
```

# 10.3.5. Relationship between change from baseline MRI scan primary endpoint (Ve, Ktrans) and change from baseline of NT-ProBNP, DLco/DLno and Ve/VCo2

Change from baseline NT-ProBNP at Scan 3 is defined as:

post constant workload exercise test –pre constant workload exercise test

The change from baseline DLco/DLno, Ve/VCo2 is defined as:

Scan 3 post MRI – Scan 3 pre-exercise

The following plots will be presented, for each component of interest as defined above:

A scatter plot, with change from baseline (Ve, Ktrans) on the horizontal axes and change from baseline NT-ProBNP, or DLco/DLno, VE/VCO2 on the vertical axes, using different colours for each population if data permit, i.e. HV and HF will be presented, as appropriate to the data.

#### 10.3.6. Analysis of Group 3 patients

For Group 3, all PD endpoints (DCE-MRI measures, lung ultrasound (B Line count), NT proBNP, dyspnoea score, and respiratory rate, etc) will be listed as appropriate. Demographic and safety (AE's if any) will still be summarized according to IDSL standards (see deliverable priority column "Group 3 SAC" for specifics in Section 12.1, note to aviod duplicated TFL numbers, all group 3 tables and listings, please add 30 into the TOC numbers. For instance for Table 9.1, use Table 9.31)

Should the following variables not being captured/calculated from the source data, they have to be calculated as followings:

LUS Score = Total line count over all zones (i.e. sum up the line counts for all zones for the subject and visit);

Inferior vena Cava Collapsability Index, IVCCI = (IVC max –IVC min)/IVC max;

Inferior vena cava diameter index, IVCDI = IVC max/ BSA

### 11. REFERENCES

European Community for Coal and Steel (ECCS), Lung Volumes and Forced Ventilatory Flows. Quanjer PH, Tammeling GJ, Cotes JE, Pedersen OF, Peslin R, Yernault J-C, 1993. 6(16):25-40.

Hankinson, JL, Odencrantz, JR, Fedan, KB. Spirometic Reference Values from a Sample of the General U.S. Population. Am J Resp Crit Care, 1999. 159:179-187.

Polgar. Pulmonary Function Testing in Children: Techniques and Standards. Philadelpahia: Sanders, 1971.

Schuirmann DJ. 1987. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability, J Pharmacokinet and Biopharm, 15, 657-680.

### 12. ATTACHMENTS

### 12.1. Table of Contents for Data Display Specifications

For the Clinical Study Report the following section numbering will apply:

Section 9: Study Population

Section 10: Safety

Section 11: Other Safety

Section 12: Efficacy

Listed below are the planned figures, tables and listings to be produced for inclusion in the MRI201137 clinical study report:

- The 'IDSL No. / Example Shell'" column refers to the relevant example in the Integrated Data Standards Library (IDSL) database
- Unless otherwise indicated, these refer to the core IDSL data standards located under:
  - o 'Data Standards' → 'By Component' in the IDSL database


# 12.2. Study Population and Disposition

# 12.2.1. Study population

### <u>Listings</u>

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming<br>Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 9.1 | Safety | IE3 | Listing of Analysis populations | | Programmer | SAC, Group 3<br>SAC |

# 12.2.2. Disposition

### <u>Tables</u>

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 9.1 | Safety | ES1 | Summary of Subject Disposition | | Programmer | SAC, Group 3<br>SAC |

### <u>Listings</u>

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 9.2 | Safety | ES2 | Listing of Reasons for Study Withdrawal | | Programmer | SAC, Group 3<br>SAC |

# 12.2.3. Demography and Baseline Characteristics

### <u>Tables</u>

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 9.2 | Safety | DM1 | Summary of Demographic Characteristics | Include all variables collected. | Programmer | SAC, Group 3<br>SAC |
| 9.3 | Safety | DM5 | Summary of Race and Racial Combinations | | Programmer | SAC |

## **Listings**

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 9.3 | Safety | DM2 | Listing of Demographic Characteristics | Include all variables collected. | Programmer | SAC, Group 3<br>SAC |
| 9.4 | Safety | DM9 | Listing of Race | | Programmer | SAC, Group 3<br>SAC |

# 12.3. Safety

# 12.3.1. Exposure to MRI

### <u>Tables</u>

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 10.1 | Safety | EX1 | Summary of Exposure to MRI | Present subjects who were exposed to 1, 2, or 3 MRI scans | Programmer | SAC |


# <u>Listings</u>

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 10.1 | Safety | EX3 | Listing of Exposure to MRI | Present all MRI data. | Programmer | SAC, Group 3<br>SAC |

# 12.3.2. Laboratory Data

# <u>Tables</u>

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 10.2 | Safety | LB1 | Summary of Laboratory Values by session and overall | Include all Laboratory values collected, by Session 0, 1, 2, 3,include immediately before and after both exercise tests | Programmer | SAC Group 3<br>SAC |
| 10.3 | Safety | LB2 | Summary of Abnormal Laboratory Values by session and overall | | Programmer | SAC |
| 10.4 | Safety | UR1 | Summary of Urinalysis Data by Session and overall | | Programmer | SAC |

# <u>Listings</u>

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 10.2 | Safety | | Listing of Laboratory Data | Include all lab values, at all-time points. | Programmer | SAC, Group 3<br>SAC |
| 10.3 | Safety | LB5 | Listing of Laboratory Data for Subjects with<br>Abnormalities of Potential Clinical Concern | Include Session variable | Programmer | SAC, Group 3<br>SAC |

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 10.4 | Safety | LB13 | Listing of Laboratory Test Reference Ranges | Include Session variable | Programmer | SAC, Group 3<br>SAC |

# 12.4. Other Safety

# 12.4.1. Vital Signs

# <u>Tables</u>

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 10.5 | Safety | VS1 | Summary of Vital Signs by Session | Include all vital signs variables collected and all time points i.e. screening, after MRI scan 1 and 2, and immediately pre and post maximal and constant workload exercise tests. | Programmer | SAC, Group 3<br>SAC |
| 10.6 | Safety | VS1 | Summary of change from pre-exercise for vital signs | | Programmer | SAC |

# Listings

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 10.5 | Safety | VS4 | Listing of Vital Signs | Include change from pre-<br>exercise and session<br>variable. | Programmer | SAC, Group 3<br>SAC |


# 12.4.2. ECG

# <u>Tables</u>

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 10.7 | Safety | EG1 | Summary of ECG findings at screening | | Programmer | SAC |
| 10.8 | Safety | EG2 | Summary of ECG values at screening | | Programmer | SAC, Group 3<br>SAC |

## <u>Listings</u>

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 10.6 | Safety | EG3 | Listing of ECG values at screening | | Programmer | SAC, Group 3<br>SAC |
| 10.7 | Safety | EG5 | Listing of ECG findings at screening | | Programmer | SAC, Group 3<br>SAC |


# 12.5. Efficacy

# 12.5.1. Primary endpoint

# <u>Tables</u>

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 11.1 | Evaluable | Example A | Analysis of contrast agent interstitial volume ( $v_e$ ) and exchange rate ( $k^{trans}$ ) data | For Total lung, Left lung,<br>Right lung, Left lung<br>apical,Left lung<br>basal,Right lung apical,<br>Right lung basal | Statistician | SAC |
| 11.2 | Safety | Example A | Analysis of contrast agent interstitial volume ( $v_e$ ) and exchange rate ( $k^{trans}$ ) data | For Total lung, Left lung,<br>Right lung, Left lung<br>apical,Left lung<br>basal,Right lung apical,<br>Right lung basal | Statistician | SAC |
| 11.3 | Evaluable | VS1 | Summary of change from baseline of contrast agent interstitial volume ( $v_e$ ) and exchange rate ( $k^{trans}$ ) data | For Total lung, Left lung,<br>Right lung, Left lung<br>apical,Left lung<br>basal,Right lung apical,<br>Right lung basal | Programmer | SAC |
## Figures

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 11.101 | Evaluable | Example B | Mean (SE) Plot of contrast interstitial volume $(v_e)$ and exchange rate $(k^{trans})$ data | For Total lung, Left lung,<br>Right lung, Left lung<br>apical,Left lung<br>basal,Right lung apical,<br>Right lung basal. Separate<br>line for HF and HV. | Programmer | SAC |

# 12.5.2. Secondary endpoint

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 11.4 | Evaluable | Example A | Analysis of within subject variability of DCE-MRI<br>measures of pulmonary edema and vascular<br>permeability | Amend footnote to: Analysis performed using mixed effect model with subject (nested within scanning session) treated as a random effect, patient population (HF or HV) and scanning session (Session 1 and 2) as fixed effects. | Statistician | SAC |

## 12.5.3. Exploratory endpoint

### 12.5.3.1. Exploratory analysis of DCE-MRI measurements: Plasma volume (v<sub>p</sub>), T<sub>1</sub> relaxation rate, proton density

### <u>Tables</u>

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 11.5 | Evaluable | DM1 | Summary of DCE-MRI measurements interstitial volume ( $v_e$ ), exchange rate ( $k^{trans}$ ) (Plasma volume ( $v_p$ ), $T_1$ relaxation rate, proton density, by visit. | Replace demographic<br>variables with Plasma<br>volume (Vp), T1 relaxation<br>rate, proton density by<br>visit. | Programmer | SAC |
| 11.6 | Evaluable | DM1 | Summary of lung ultrasound total B-line scores by visit. | Replace demographic variables with LUS B-line total scores (counts). | Programmer | |

#### <u>Figures</u>

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 11.102 | Evaluable | Example B | Mean (SE) Plot for DCE-MRI measure interstitial volume $(v_e)$ . | For Total lung, Left lung, Right lung, Left lung apical,Left lung basal,Right lung apical, Right lung basal. Separate line for HF and HV patients across 3 scans. | Programmer | SAC |
| 11.103 | Evaluable | Example B | Mean (SE) Plot for DCE-MRI measure exchange rate (k <sup>trans</sup> ) | For Total lung, Left lung, Right lung, Left lung apical, Left lung basal, Right lung apical, Right lung basal. Separate line for HF and HV patients across 3 scans. | Programmer | SAC |

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 11.104 | Evaluable | Example B | Mean (SE) Plot for DCE-MRI measure Plasma volume (v <sub>p</sub> ). | For Total lung, Left lung, Right lung, Left lung apical, Left lung basal, Right lung apical, Right lung basal. Separate line for HF and HV patients across 3 scans. | Programmer | SAC |
| 11.105 | Evaluable | Example B | Mean (SE) Plot for DCE-MRI measure T <sub>1</sub> relaxation rate. | For Total lung, Left lung, Right lung, Left lung apical, Left lung basal, Right lung apical, Right lung basal. Separate line for HF and HV patients across 3 scans. | Programmer | SAC |
| 11.106 | Evaluable | Example B | Mean (SE) Plot for DCE-MRI measure proton density. | For Total lung, Left lung, Right lung, Left lung apical, Left lung basal, Right lung apical, Right lung basal. Separate line for HF and HV patients across 3 scans. | Programmer | SAC |
| 11.201 | Evaluable | Example C | Spaghetti plot of interstitial volume (v <sub>e</sub> ) by scan session | For Total lung, Left lung, Right lung, Left lung apical, Left lung basal, Right lung apical, Right lung basal. Interstitial volume (Ve) on the vertical axes, scan session on the horizontal axes, and different symbols for HF and HV patients. (3 Scans) | Programmer | SAC |
| 11.202 | Evaluable | Example C | Spaghetti plot of exchange rate (k <sup>trans</sup> ) by scan session | For Total lung, Left lung, Right lung, Left lung apical, Left lung basal, Right lung apical, Right lung basal. Exchange rate (k <sup>trans</sup> ) on the vertical axes, scan session on the horizontal axes, and different symbols for HF and HV patients. | Programmer | SAC |
| 11.301 | Evaluables | Example D | Scatter plot of change from baseline interstitial volume (v <sub>e</sub> ) and change from baseline Pro-BNP | | Programmer | SAC |

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 11.302 | Evaluables | Example D | Scatter plot of change from baseline interstitial volume (ve) and change from baseline DLno/DLco | | Programmer | SAC |
| 11.303 | Evaluables | Example D | Scatter plot of change from baseline interstitial volume (v <sub>e</sub> ) and change from baseline Ve/VCo2 | | Programmer | SAC |
| 11.304 | Evaluables | Example D | Scatter plot of<br>change from<br>baseline exchange<br>rate (k <sup>trans</sup> ) and<br>Change from<br>baseline Pro-BNP | | Programmer | SAC |
| 11.305 | Evaluables | Example D | Scatter plot of change from baseline exchange rate (k <sup>trans</sup> ) and Change from baseline DLno/DLco | | Programmer | SAC |

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 11.306 | Evaluables | Example D | Scatter plot of change from baseline exchange rate (k <sup>trans</sup> ) and Change from baseline Ve/VCo2 | | Programmer | SAC |

## 12.5.3.2. Comparison of DLco/DLno gas diffusion parameters at baseline by group (HF, HV)

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 11.6 | Evaluable | DM1 | Summary of gas diffusion, lung function parameters by visit. | | Programmer | SAC |
| 11.7 | Evaluable | Example A | Analysis of gas diffusion parameters: parameters DLno, DLco, and DLno/DLco ratio at baseline. | Using mixed model to compare all parameters of interest between HF and HV if data permit. | Statistician | SAC |

#### **Figures**

| 11.401 | Evaluable | Example B | Mean (SE) Plot for gas<br>diffusion (DLno, DLco and<br>DLco/DLno) , lung<br>function parameter | Separate line for HF and HV patients across 3 scans, a separate plot for each gas diffusion, lung function parameter | Programmer | SAC |
|---|---|---|---|---|---|---|
| 11.501 | Evaluable | Example C | Spaghetti plot of gas<br>diffusion parameter by<br>scan session (DLno, DLco<br>and DLco/DLno) | Gas diffusion parameter on the vertical axes, scan session on the horizontal axes, and different symbols for HF and HV patients, a separate plot for each gas diffusion parameter | Programmer | SAC |

### 12.5.3.3. Comparison of Dyspnoea Score at baseline by group (HV, HF)

### <u>Tables</u>

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 11.8 | Evaluable | DM1 | Summary of Dyspnoea score by visit and session | Use dyspnoea variables at each planned time point, including immediately before and after both exercise tests. | Programmer | SAC |

### **Figures**

| 11.6 | Evaluable Example F | Frequency bar plot of Dyspnoea score by visit | Programmer | SAC |
|---|---|---|---|---|
|---|---|---|---|---|

#### 12.5.3.4. Comparison of Respiratory Rate at baseline by group (HV, HF)

#### <u>Tables</u>

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 11.9 | Evaluable | DM1 | Summary of Respiratory rate by visit | Use respiratory rate at each planned time point. | Programmer | SAC |

#### **Figures**

| 11.7 | Evaluable | Example B | Mean (SE) Plot for respiratory rate by visit. | Separate line for HF and HV patients across 3 | Programmer | SAC |
|---|---|---|---|---|---|---|
| | | | | scans. | | |

### 12.5.3.5. Comparison of effect of exercise at Scan 3 by group (HV, HF)

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 11.10 | Evaluable | Example A | Analysis of effect of exercise (session 3) on gas diffusion parameters | Amend footnote to: Analysis performed using a mixed effect model, subject is random effect, (HF or HV) as fixed effects. With change from pre-exercise gas diffusion parameters DLno, DMco, for both exercise tests. | Statistician | SAC |

## 12.5.3.6. Comparison of exercise test parameters at Scan 3 by group (HV, HF)

| No. | Population | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 11.11 | Evaluable | DM1 | Summary of exercise test parameters | Use the data collected at scan 3, no pre/post or change from baseline values. | Programmer | SAC |
| 11.12 | Evaluable | Example A | Analysis of exercise test parameters of interest (Ve/Vco2 ratio at Scan 3 by HF and HV. | Use the data collected at scan 3, no pre/post or change from baseline values. | Statistician | SAC |

#### 12.5.3.7. Relationship between exercise parameters (Ve/Vco2) vs gas diffusion DLno/DLco parameters at scan 3

#### <u>Listings</u>

| No. | Population <sup>1</sup> | IDSL No. /<br>Example Shell | Title | Additional Programming Notes | Responsibility | Deliverable<br>Priority |
|---|---|---|---|---|---|---|
| 11.1 | 1.1 Evalauble | | Listing of DCE-MRI scan data | | Programmer | SAC. Group 3<br>SAC |
| 11.2 | Evalauble Listing of dyspnoea score | | Include all variables collected. | Programmer | SAC, Group 3<br>SAC | |
| 11.3 | Evalauble | | Listing of respiratory rate | Include all variables collected. | Programmer | SAC, Group 3<br>SAC |
| 11.4 | Evalauble L | | Listing of NT-proBNP measurements | -proBNP measurements Include all variables collected. | | SAC, Group 3<br>SAC |
| 11.5 | Evalauble | Listing of exercise capacity measuren | | Include all variables collected. | Programmer | SAC, Group 3<br>SAC |
| 11.6 | Evalauble | Listing of DLco and DLno measurements | | Include all variables collected. | Programmer | SAC, Group 3<br>SAC |
| 11.7 | 11.7 Evalauble | | Listing of plasma volume $(v_p)$ | Include all variables collected. | Programmer | SAC, Group 3<br>SAC |
| 11.8 | Evalauble | | Listing of T <sub>1</sub> relaxation rate and proton density | Include all variables collected. | Programmer | SAC |
| 11.7 | Evalauble | | Listing of Lung Ultrasound Data and Score | Include all variables collected, including B-line counts, total scores as well as by thoracic zones | Programmer | Group 3 SAC |

<sup>&</sup>lt;sup>1</sup> Evaluable population is not applicable to Group 3, using Safety population for Group 3 displays

#### 12.6. Data Display Specifications (Example Shells)

Example : Example A Page 1 of n

Protocol : 2013N186309\_02

Population : Completers

#### Table X.X

Analysis of contrast agent interstitial volume ( $v_e$ ) and exchange rate ( $k^{trans}$ ) data for total lung, left lung, right lung, left apical segments, right apical segment and left basal segment

Pls update this mock table with headers something as the following:

| | | Comparisons (C | Grp1 vs Grp0) | LSMean | (Se) | Point estimate | es |
|---|---|---|---|---|---|---|---|
| Parameter | Region | Group1 | Group0 | Group1 | Group0 | and 95% CI | p-value |
| Ve | Left<br>Lung | HF (n=) Post Exercise | HV (n=) Session 2 | xxx.xx(xx.x) | xxx.xx(xx.xx) | xx.xx(xx.xx,<br>xx.xx) | 0.xx |
| | | in HF (n=) | in HF (n=) | xxx.xx(xx.x) | xxx.xx(xx.xx) | xx.xx(xx.xx,<br>xx.xx) | 0.xx |


Example : Example A (Secondary Objective)

Protocol: 201137 Page 1 of 6

Population: Evaluable

Table 11.3

Analysis of within subject variability of DCE-MRI measures of pulmonary edema

and vascular permeability

Comparisons: (Session 2 Vs Session 1)

| MRI | Region<br>of | | GeoMean ( | Se in log) | Point estimates | | of Variat<br> | |
|---|---|---|---|---|---|---|---|---|
| | | | Session2 | Session1 | (Ratio) and 95% CI | p-value | by pop | |
| Transfer rate from | Lungs | Heart Failure<br>(n=12) | 0.187<br>(0.129) | 0.206<br>(0.193) | 0.908<br>(0.634, 1.300) | 0.5789 | 32.4 | 43.3 |

plasma to extracellu lar space (EES) (Ktrans) (1/MIN)

Example : Example B

Protocol : 2013N186309 02

Population : Completers


#### Figure *X.X*

Mean (SE) Plot, Analysis performed using a Mixed effect model with subject (nested within scanning session) treated as a random effect, patient population (HF or HV) and Scanning Session (Session 1 and 2) as fixed



effects

Example : Example C

Protocol : 2013N186309 02

Population : Completers

48

Figure X.X



Example Protocol

: Example D : 2013N186309\_02 : Completers

Population


Figure X.X

#### ApoA1 CH (%) at week 8 vs. Baseline NEFA (MEQ/L)



Amend title to "Scatter plot of var 1 vs var 2. Amend axes labels to appropriate variable names Amend legend text to Healthy Volunteers and Heart Failure patients.

Example: Example E
Protocol: 2013N186309\_02
Population: Completers


 $\hbox{Table xx.xx}$  Correlation of Change from Baseline in MRI Parameters and Change from Baseline NT-proBNP Analysis

| | Parameter 1 | Parameter 2 | Group | Pearson's<br>Correlation (P-<br>value) | Spearman's<br>Correlation (P-value) |
|---|---|---|---|---|---|
| Left Lung | | | | | |
| Apical segment | MRI Parameter | NT-proBNP<br>Parameter | Healthy volunteers | x.xxxx (0.xxxx) | x.xxxx (0.xxxx) |
| | MRI Parameter | NT-proBNP<br>Parameter | Heart failure | x.xxxx (0.xxxx) | x.xxxx (0.xxxx) |
| Basal<br>segment | MRI Parameter | NT-proBNP<br>Parameter | Healthy volunteers | x.xxxx (0.xxxx) | x.xxxx (0.xxxx) |
| | MRI Parameter | NT-proBNP<br>Parameter | Heart failure | x.xxxx (0.xxxx) | x.xxxx (0.xxxx) |
| Total | MRI Parameter | NT-proBNP<br>Parameter | Healthy<br>volunteers | x.xxxx (0.xxxx) | x.xxxx (0.xxxx) |
| | MRI Parameter | NT-proBNP<br>Parameter | Heart failure | x.xxxx (0.xxxx) | x.xxxx (0.xxxx) |
| Right Lung | | | | | |

| Apical segment | MRI Parameter | NT-proBNP<br>Parameter | Healthy volunteers | x.xxxx (0.xxxx) | x.xxxx (0.xxxx) |
|---|---|---|---|---|---|
| | MRI Parameter | NT-proBNP<br>Parameter | Heart failure | x.xxxx (0.xxxx) | x.xxxx (0.xxxx) |
| Basal<br>segment | MRI Parameter | NT-proBNP<br>Parameter | Healthy volunteers | x.xxxx (0.xxxx) | x.xxxx (0.xxxx) |
| | MRI Parameter | NT-proBNP<br>Parameter | Heart failure | x.xxxx (0.xxxx) | x.xxxx (0.xxxx) |
| Total | MRI Parameter | NT-proBNP<br>Parameter | Healthy volunteers | x.xxxx (0.xxxx) | x.xxxx (0.xxxx) |
| | MRI Parameter | NT-proBNP<br>Parameter | Heart failure | x.xxxx (0.xxxx) | x.xxxx (0.xxxx) |
| Total both lungs | MRI Parameter | NT-proBNP<br>Parameter | Healthy volunteers | x.xxxx (0.xxxx) | x.xxxx (0.xxxx) |
| | MRI Parameter | NT-proBNP<br>Parameter | Heart failure | x.xxxx (0.xxxx) | x.xxxx (0.xxxx) |

Example : Example D Page 1 of n
Protocol : 2013N186309\_02

Protocol : 2013N186309\_02 Population : Evaluable

Frequency bar plot of Dyspnoea score by visit

